CLINICAL TRIAL: NCT06507436
Title: The Efficacy and Safety of Herombopag in Treating Thrombocytopenia in Chronic Liver Disease Patients Undergoing Elective Invasive Surgery - A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study
Brief Title: The Phase III Clinical Study of Herombopag for the Treatment of Thrombocytopenia in Chronic Liver Disease Patients Undergoing Elective Invasive Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8735-302
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Thrombocytopenia in Chronic Liver Disease Patients Undergoing Elective Invasive Surgery

STUDY DESIGN:
Intervention Model Description: Herombopag compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group 1 (Experimental)
  Interventions: Drug: Herombopag tablets; Drug: Herombopag placebo tablets
- Treatment group 2 (Experimental)
  Interventions: Drug: Herombopag tablets; Drug: Herombopag placebo tablets

INTERVENTIONS:
Drug: Herombopag tablets — Herombopag tablets; dose 1 or dose 2, for 5 days
Drug: Herombopag placebo tablets — Herombopag placebo tablets; dose 1 or dose 2, for 5 days

SUMMARY:
This study includes Part A and Part B. Part A is a dose-finding study for subjects with chronic liver disease-related thrombocytopenia scheduled for elective surgery. Part B is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study designed to evaluate the efficacy and safety of Herombopag compared to placebo in patients with chronic liver disease-related thrombocytopenia undergoing elective invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 years or older withc a Child-Pugh score of Class A or Class B;
2. Platelet count less than 50×10^9/L on baseline;
3. Elective invasive procedures or surgeries that are planned.

Exclusion Criteria:

1. Any history of arterial or venous thrombosis, including partial or complete thrombosis;
2. Evidence of thrombosis (partial or complete) in the main portal vein, portal vein branches, or any part of the splenic mesenteric system at Screening;
3. Portal vein blood flow velocity rate <10 centimeters/second at Screening;
4. There are other diseases that may cause thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Part A: CL/F | 0 minute to 5 days
Part A: Vc/F | 0 minute to 5 days
Part A: ka | 0 minute to 5 days
Part A: Q/F | 0 minute to 5 days
Part A: AUC0-tau | 0 minute to 5 days
Part A: Cmax | 0 minute to 5 days
Part A: Kin | 0 minute to 35 days
Part A: Kout | 0 minute to 35 days
Part A: Kdeg | 0 minute to 35 days
Part A: Slope | 0 minute to 35 days
The proportion of subjects whose platelet count is ≥50×10^9/L within 24 hours before surgery and has increased by ≥20×10^9/L from baseline, and who have not received platelet transfusion or other treatments to raise platelet levels before surgery | 0 minute to 11 days
  Part B

SECONDARY OUTCOMES:
The proportion of subjects with a platelet count of ≥50×10^9/L within 24 hours before surgery | 0 minute to 11 days
The duration of time during the study when the platelet count remains ≥50×10^9/L | 0 minute to 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, affiliated with Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided